

« Etude sur l'observation de l'évolution des symptômes sexuels chez les délinquants sexuels atteints de paraphilie (avec ou sans traitements antiandrogènes ou ISRS) »
- ESPARA -

Cette recherche est organisée par le Groupe Hospitalier Universitaire – Psychiatrie et neurosciences (GHU Paris) Délégation à la Recherche Clinique et à l'Innovation (DRCI) 1, rue Cabanis 75014 Paris

#### NOTE D'INFORMATION ET CONSENTEMENT PATIENT

Madame, Monsieur,

Il est important de lire attentivement cette note avant de prendre votre décision ; n'hésitez pas à lui demander des explications. Vous pouvez prendre un temps de réflexion jusqu'à 7 jours (maximum) pour lire les renseignements qui suivent.

Si vous décidez de participer à cette recherche, un consentement écrit vous sera demandé. Si vous choisissez de ne pas prendre part à l'étude, ceci n'aura aucune conséquence sur votre prise en charge médicale.

#### 1) Introduction

Jusqu'à présent, peu d'études menées sur des petites séries de patients ont été publiées et les connaissances scientifiques sur le traitement des délinquants sexuels paraphiles sont modestes.

Les traitements médicamenteux actuellement utilisés dans la prise en charge des paraphilies sont :

- les inhibiteurs de la recapture de la sérotonine (ISRS),
- et les anti androgènes.

En fonction de la gravité de la paraphilie, l'un et/ou l'autre ou aucun des deux peuvent être utilisés (selon les recommandations nationales de la Haute Autorité de Santé et internationales de la World Federation of Societies of Biological Psychiatry (WFSBP)). Afin de mieux connaître l'efficacité et les effets secondaires de ces médicaments, nous vous proposons de participer à cette étude, au cours de laquelle votre prise en charge médicale et psychologique ne sera pas modifiée.

## 2) Quel est le but de cette recherche?

L'objectif de cette recherche, à laquelle nous vous proposons de participer est d'évaluer les symptômes sexuels chez les sujets paraphiles inclus dans l'étude (3 groupes de patients : patients sous antiandrogènes, patients sous les inhibiteurs de la recapture de la sérotonine (ISRS) et patients sans traitements pharmacologiques de types ISRS ou antiandrogène).



## 3) En quoi consiste cette recherche?

Les objectifs de cette étude sont non seulement de mieux connaître le profil des personnes bénéficiant ou non d'un traitement médicamenteux dans la prise en charge de la paraphilie\* (données socio-économiques, histoire de vie notamment traumatique, types de soins reçus, maladies somatiques associées (diabète, hypertension artérielle,...), addictologique (consommation de tabac, alcool, drogues...), psychiatrique (anxiété, dépression...)...) mais surtout de pouvoir étudier l'efficacité, le retentissement sur la qualité de vie des traitements reçus. Elle permettra également de mieux étudier les effets secondaires de ces traitements.

Pour répondre à la question posée dans la recherche, il est prévu d'inclure 200 personnes ayant commis un délit ou une agression sexuelle et présentant une paraphilie, dans des établissements de soins situés dans différents centres en France.

## 4) Quel est le calendrier de la recherche?

La durée prévisionnelle du projet de recherche (inclusion et suivi) est de 5 ans et votre participation durera 3 ans.

#### 5) Comment va se dérouler cette étude ?

Après la signature de votre consentement, lors de la première visite, le déroulement de la recherche sera le suivant :

Après des explications générales sur le contexte de l'étude et après avoir répondu à toutes vos questions, l'investigateur confirmera auprès de vous l'absence de critères de non inclusion et recueillera votre accord écrit pour participer à cette étude.

Lors de votre première visite, les informations suivantes seront recueillies par autoquestionnaires ou lors d'un entretien avec le médecin ou une infirmière formée pour cette étude : données socioéconomiques, antécédents personnels et familiaux (somatiques, addictologiques, psychiatriques, sexuels), histoire de vie, parcours de soin et parcours juridique, données sur le comportement sexuel (fantasmes, activités sexuelles).

\*Paraphilie: comportements sexuels comme pédophilie, exhibitionnisme, sadisme sexuel...

Des questionnaires vous seront proposés : recherche de trouble psychiatrique, évaluation de la personnalité, recherche de psychotraumatisme et impact d'un traumatisme notamment sexuel, évaluation cognitive, échelle de dépression, échelle d'idéation suicidaire, échelle afin de rechercher et d'évaluer une hypersexualité éventuelle, échelle de désir et intensité sexuelle, échelle de qualité de vie et échelles d'évaluation cognitive. La durée de passation des tests et échelles lors de la première visite sera d'environ quatre heures.



Un bilan biologique sera également réalisé à l'inclusion. Enfin, une mesure de votre densité osseuse sera réalisée à l'inclusion et en fin d'étude (3 ans après votre inclusion) (seulement si vous prenez des antiandrogènes ou des ISRS).

<u>Un suivi tous les trois mois</u> vous sera ensuite proposé sur une durée de 36 mois. A chaque séance seront recueillis les évènements de vie intercurrents\*, des éléments sur la tolérance et l'efficacité du traitement si vous en avez un, la recherche d'effets indésirables du traitement s'il y a lieu. La durée de la passation des tests et questionnaires sera environ d'une heure par visite.

\* Intercurrents : évènements qui surviennent au cours d'une autre maladie (Rechute, usage d'alcool et de drogues illicites...etc.)

<u>Lors de la dernière visite</u> prévue 3 ans après votre inclusion, une visite semblable à la visite d'inclusion sera réalisée.

## 6) Prélèvements biologiques

Un prélèvement de salive et un prélèvement sanguin seront également réalisés le jour de votre <u>inclusion</u>. Ces prélèvements sont réalisés pour des analyses génétiques.

## 7) Quels sont les bénéfices liés à votre participation ?

Il n'y aura pas de bénéfice direct pour vous, mais votre participation contribuera à améliorer les connaissances sur les indications de ces traitements, qui pourraient éventuellement être revues en ce qui concerne leur efficacité et la tolérance.

## 8) Quels sont les risques et les contraintes liés à la recherche?

8.1 Contraintes

Si vous acceptez de participer, vous devrez respecter les points suivants :

- Conserver sur vous en permanence la carte patient qui vous a été remise, indiquant que vous participez à cette recherche. Cette carte inclut le nom et le numéro de téléphone de votre médecin,
- Venir aux rendez-vous prévus dans le cadre de votre suivi. En cas d'impossibilité, nous vous remercions de contacter votre médecin le plus rapidement possible.
- Informer le médecin de la recherche de l'utilisation de tout médicament ainsi que de tout événement survenant pendant la recherche (hospitalisation, ...),
- Le médecin investigateur peut arrêter ma participation à l'étude (la raison de cet arrêt sera expliquée)
- Ne pas prendre part à un autre projet de recherche sans l'accord de votre médecin,
- Être affilié(e) à un régime de sécurité sociale ou être bénéficiaire d'un tel régime.



## 8.2 Risques

L'examen de la mesure de la densité osseuse fait partie des examens complémentaires envisagés lors d'un suivi classique (<u>seulement si vous prenez des antiandrogènes</u>) et le risque de cet examen est très faible.

#### 9) Remboursement des frais et indemnisation

Votre participation à cette recherche n'entrainera pas de participation financière de votre part, autre que celle liée à votre prise en charge habituelle. Tous les frais liés à cette recherche sont à la charge du promoteur.

Aucune indemnisation n'est prévue pour les patients se prêtant à la recherche.

# 10) Si vous acceptez de participer, que vont devenir vos données recueillies pour la recherche ?

Ces données ne seront pas transmises à un pays hors de l'Union Européenne ou à une organisation internationale. Ces données resteront sur le territoire national.

Vous pouvez retirer à tout moment votre consentement à l'utilisation ultérieure de vos données auprès du médecin qui vous suit dans le cadre de cette recherche. Pour tout arrêt de participation au cours de l'étude, les données recueillies précédemment à cet arrêt seront utilisées conformément à la réglementation.

- Données identifiantes : Les informations concernant votre identité (nom, prénom) ne seront connues que par l'équipe médicale vous prenant en charge ainsi que par les personnes réalisant le contrôle de la qualité de la recherche et mandatées par le promoteur. Le cas échéant, ces données pourront être accessibles aux autorités sanitaires ou de contrôle, au délégué à la protection des données du promoteur si vous le contactez et, en cas de litige, par le personnel habilité de l'organisme d'assurance du promoteur. Ces personnes sont soumises au secret professionnel.
- Données pseudonymisées : Les données seront collectées dans la mesure où elles sont nécessaires à la recherche : histoire de la maladie, traitements reçus, antécédents médicaux, paramètres vitaux, ECG, examens biologiques. Les données recueillies seront traitées de manière confidentielle, conformément à la loi du 6 janvier 1978 modifiée dite « Loi Informatique et Libertés », et au Règlement Général sur la Protection des Données (RGPD).

Vos données seront pseudonymisées, c'est-à-dire identifiées par un numéro de code, sans mention de vos noms et prénoms.

Vos données pseudonymisées seront accessibles au promoteur GHU Psychiatrie et Neurosciences et aux personnes agissant pour son compte.

Ces personnes, soumises au secret professionnel, auront accès à vos données pseudonymisées dans le cadre de leur fonction et en conformité avec la réglementation. Vos données pseudonymisées seront conservées en base active le temps nécessaire à leur analyse et à la publication des résultats,



puis archivées conformément à la réglementation en vigueur pendant 15 ans. La publication des résultats de l'étude ne comportera aucun résultat individuel.

## 11) Que vont devenir vos échantillons recueillis à la fin de la recherche?

Les échantillons issus des prélèvements sanguins et salivaires réalisés dans le cadre de la recherche feront l'objet de collections biologiques, en vue de recherches ultérieures. Ces échantillons ne feront pas l'objet d'analyses pendant la recherche.

Au cours de la recherche, ces échantillons destinés aux collections biologiques seront centralisés et conservés à l'institut de Psychiatrie et Neurosciences à Paris (unité INSERM U 1266) sous la responsabilité du Pr THIBAUT.

L'échantillon salivaire se conserve à température ambiante et les prélèvements sanguins (deux tubes EDTA 4ml de sang) sont stockés dans un congélateur (entre -20° et -80° C).

Les échantillons biologiques conservés pourront faire l'objet de recherche génétiques futures sur une meilleure compréhension des comportements à l'origine des délits sexuels.

Ces échantillons pourront également être utilisés pour des analyses ultérieures non prévues dans le protocole pouvant se révéler intéressantes dans le cadre de la pathologie, en fonction de l'évolution des connaissances scientifiques, sous réserve que vous n'y soyez pas opposé. Les prélèvements restants non utilisés lors des analyses seront systématiquement détruits. A la fin de la recherche, ces collections biologiques seront déclarées auprès du ministère chargé de la recherche. »

Vous avez la possibilité à tout moment de demander au médecin qui vous suit dans le cadre de la recherche, la destruction de ces prélèvements biologiques ou de vous opposer à toute utilisation ultérieure.

#### 12) Comment cette recherche est-elle encadrée?

Le GHU Paris - Psychiatrie et Neurosciences, promoteur de la recherche, a pris toutes les mesures pour mener cette recherche conformément aux dispositions du Code de la Santé Publique applicables aux recherches impliquant la personne humaine.

Cette recherche entre dans le cadre de la « Méthodologie de Référence pour les traitements de données personnelles opérés dans le cadre des recherches impliquant la personne humaine » (MR-001). Le GHU - Paris Psychiatrie et Neurosciences a signé un engagement de conformité à cette « Méthodologie de Référence »

Le GHU Paris - Psychiatrie et Neurosciences a souscrit une assurance (n° de police 163543) garantissant sa responsabilité civile et celle de tout intervenant auprès de la compagnie Relyens Mutual Insurance dont l'adresse est 18 rue Edouard Rochet 69372 LYON cedex 08, comme prévu à l'article L1121-10 du Code de la Santé Publique.

Le GHU Paris - Psychiatrie et Neurosciences a obtenu l'avis favorable du Comité de Protection des Personnes (CPP) Est IV pour la réalisation de cette recherche le 20/03/2025.



Le GHU Paris - Psychiatrie et Neurosciences, promoteur, transmettra, pour information à l'ANSM, l'avis favorable du CPP et le résumé du protocole.

Conformément à la réglementation en vigueur, pour participer à cette recherche vous devez être affilié(e) à un régime de sécurité sociale.

A l'issue de la recherche et après analyse des données relatives à cette étude, vous pourrez être informé(e) des résultats globaux par l'intermédiaire du médecin vous ayant proposé de participer à la recherche.

#### 13) Quels sont vos droits?

Conformément aux dispositions de la loi n° 78-17 du 6 janvier 1978 modifiée relative à l'informatique, aux fichiers et aux libertés et au Règlement Général sur la Protection des Données (RGPD - Règlement (UE) 2016/679), vous disposez d'un droit d'accès et de rectification, d'un droit à l'effacement (droit à l'oubli) et d'un droit à la limitation du traitement de vos données. Vous pouvez également accéder directement ou par l'intermédiaire d'un médecin de votre choix à l'ensemble de vos données médicales en application des dispositions de l'article L.1111-7 du Code de la Santé Publique. Vous disposez également d'un droit d'opposition, à tout moment, à l'utilisation et/ou à la transmission des données couvertes par le secret professionnel susceptibles d'être utilisées dans le cadre de cette recherche et d'être traitées. Vous pouvez renoncer à tout moment à participer à la recherche sans avoir à vous justifier. Sachez toutefois que les données recueillies préalablement au retrait de votre participation, à l'exercice de votre droit à l'effacement ou à l'exercice de votre droit d'opposition pourraient ne pas être effacées si leur effacement risque de rendre impossible ou de compromettre la réalisation des objectifs de la recherche.

Le promoteur n'ayant pas accès à votre identité, ces droits s'exercent dans un premier temps auprès du médecin investigateur qui vous suit dans le cadre de cette recherche.

Pour toute question relative à la protection des données ou pour exercer vos droits, vous pouvez contacter le délégué à la protection des données désigné par le promoteur à l'adresse suivante : dpo@ghu-paris.fr ou par voie postale avec la mention à l'attention du DPO du GHU Paris - Psychiatrie et Neurosciences, 1 rue Cabanis, 75674 Paris Cedex 14.

Dans le cas vous contactez le DPO votre anonymat sera levé mais le DPO est soumis au secret professionnel

Conformément à l'article 77 du RGPD, vous avez le droit d'introduire une réclamation auprès de la Commission nationale de l'informatique et des libertés (CNIL), si vous considérez que le traitement de vos données n'est pas en conformité avec ledit règlement, directement en ligne (https://www.cnil.fr/fr/plaintes) ou par courrier postal à l'adresse : CNIL – Service des Plaintes – 3



Place de Fontenoy – TSA 80715 – 75334 PARIS CEDEX 07. La CNIL est l'autorité de contrôle compétente en France en matière de protection des données.

# 14) Libre choix de participation

Votre participation à cette recherche est entièrement libre et volontaire. Vous pouvez vous retirer à tout moment de la recherche sans justification. Cela n'entraînera aucun préjudice ni changement dans votre prise en charge habituelle.

Vous pourrez tout au long de la recherche demander des explications sur le déroulement de la recherche au médecin investigateur.

Si vous acceptez de participer à la recherche après avoir lu toutes ces informations et discuté tous les aspects avec le médecin en charge de la recherche, vous devrez signer et dater le formulaire de consentement éclairé se trouvant à la fin de ce document.



#### FORMULAIRE DE CONSENTEMENT

| Je | soussigné(e), | Mme, | M. | [rayer | les | mentions | inutiles] | (nom, | prénom) |
|---|---|---|---|---|---|---|---|---|---|
| | pte librement de<br>ptômes sexuels o | | | | | | | | |
| - | androgènes ou l | | - | | | | • | | |
| | rosciences, (GHU<br>om, téléphor | , | 1 | | 1 | | | | • |
| inve | stigateur dans ce | tte recherc | he. | | | | | | |

- J'ai pris connaissance de la note d'information version 2.0 du 07/02/2025 (07 pages) m'expliquant l'objectif de cette recherche, la façon dont elle va être réalisée et ce que ma participation va impliquer,
- Je conserverai un exemplaire de la note d'information et du consentement,
- J'ai reçu des réponses adaptées à toutes mes questions,
- J'ai disposé d'un temps suffisant pour prendre ma décision,
- J'ai compris que ma participation est libre et que je pourrai interrompre ma participation à tout moment, sans avoir à en justifier les raisons. Cela n'aura aucune conséquence sur la qualité des soins que je recevrai,
- Je suis conscient que ma participation pourra aussi être interrompue par le médecin si besoin, il m'en expliquera les raisons,
- J'ai compris que pour pouvoir participer à cette recherche je dois être affilié à un régime de sécurité sociale ou bénéficiaire d'un tel régime. Je confirme que c'est le cas,
- J'ai la possibilité de venir pour les rendez-vous accompagné par une personne de confiance,
- J'ai bien compris qu'aucune indemnité n'était prévue pour ma participation à cette recherche,
- J'ai bien noté que je dispose d'un droit d'accès, de rectification, de limitation et, le cas échéant, d'opposition et d'effacement, concernant le traitement de mes données personnelles. Ces droits s'exercent en premier lieu auprès de l'investigateur qui me suit dans le cadre de cette recherche et qui connaît mon identité,
- A l'issue de la recherche, je pourrai être informé des résultats globaux par l'intermédiaire du médecin investigateur,
- J'ai bien été informé que mes données pseudonymisées, recueillies dans le cadre de la recherche, pourront être réutilisées et partagées pour des recherches ultérieures à des fins scientifiques sauf si je m'y oppose, et que je pourrai revenir sur ma décision et m'y opposer à tout moment,



- Mon consentement ne décharge en rien le médecin qui me suit dans le cadre de la recherche ni le GHU Paris - Psychiatrie et Neurosciences de l'ensemble de leurs responsabilités, et je conserve tous mes droits garantis par la loi.
- J'ai été informé des risques et contraintes liés à ma participation au protocole »,
- J'ai été informé que le promoteur a souscrit une assurance responsabilité civile »
- J'ai été informé que mes données personnelles étaient sécurisées ».

| Signature de la personne participant à la recherche: | Signature du médecin : |
|---|---|
| Nom Prénom : | |
| | Nom Prénom : |
| Date : | Date : |
| Signature : | Signature: |

Ce document est à réaliser en 3 exemplaires, un exemplaire doit être conservé 15 ans par l'investigateur, le deuxième remis à la personne donnant son consentement et le troisième transmis au GHU Paris Psychiatrie et Neurosciences sous enveloppe scellée à la fin de la recherche.



| Consentement spécifique pour l'analyse génétique | | | | |
|---|---|---|---|---|
| J'accepte la réalisation de prélèvements dans le cadre de cette recherche. | | | | |
| Oui 🗆 | | Non [ | ☐ [coo | cher la case] |
| J'accepte que mes échantillons intègrent une collection utilisée pour des recherches futures. | | | | |
| Oui 🗆 | | Non | | [cocher la case] |
| J'accepte que mes échantillons servent à des analyses génétiques. | | | | |
| Oui 🗆 | Non 🗆 | [coch | ier la c | case] |
| J'accepte que les données enregistrées à l'occasion de cette recherche comportant des données génétiques puissent faire l'objet d'un traitement informatisé par le promoteur ou pour son compte. J'ai bien noté que le droit d'accès prévu par la loi (Loi 78-17 du 06 janvier 1978 modifiée par l'ordonnance du 12 décembre 2018) relative à l'informatique, aux fichiers et aux libertés s'exerce à tout moment auprès du médecin qui me suit dans le cadre de la recherche et qui connaît mon identité. Je pourrai exercer mon droit de rectification et d'opposition en contactant directement le DPO du GHU Paris - Psychiatrie et Neurosciences (cf. point 13 de la présente note pour ses coordonnées). | | | | |
| Oui 🗆 | | Non | □ [cc | ocher la case] |
| Signature de la personne participant à la rech | nerche | Siş | gnatui | re du médecin |
| Nom Prénom : | | No | om Pré | énom : |
| Date : | | Da | ite : | |
| Signature : | | Sig | gnatur | e : |

Ce document est à réaliser en 3 exemplaires, un exemplaire doit être conservé 15 ans par l'investigateur, le deuxième remis à la personne donnant son consentement et le troisième transmis au GHU Paris Psychiatrie et Neurosciences sous enveloppe scellée à la fin de la recherche.